CLINICAL TRIAL: NCT05443789
Title: Boosting General Practice pRescription by Individual Educational Fast Academic Detailing Visits About Proton Pump Inhibitor
Brief Title: Academic Detailing About Proton Pump Inhibitors
Acronym: BRIEF-PI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jón Þór Trærup Andersen (Other)
Responsible Party: Sponsor-Investigator, Jón Þór Trærup Andersen, Clinical Professor, University Hospital Bispebjerg and Frederiksberg
Organization: University Hospital Bispebjerg and Frederiksberg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: P-2021-709b
Record Dates: First submitted 2021-10-06; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Prescription Pattern

STUDY DESIGN:
Intervention Model Description: randomized placebo controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proton pump inhibitor education (Experimental): The general practices in this arm will receive the education visits about Proton pump inhibitor.
  Interventions: Behavioral: Proton pump inhibitor education
- Other education (Placebo Comparator): The general practices in this arm will receive an educational visit on another topic (asthma).
  Interventions: Behavioral: Other education

INTERVENTIONS:
Behavioral: Proton pump inhibitor education — A 15 minutes (preferable) one-on-one educational visit about deprescription of proton pump inhibitor
  Arms: Proton pump inhibitor education
Behavioral: Other education — A 15 minutes (preferable) one-on-one educational visit about another topic (NOT asthma).
  Arms: Other education

SUMMARY:
General practices in the Capital Region of Denmark are offered a short educational visit and are randomized to either proton pump inhibitor (intervention) or another topic (control).

The change in prescription pattern from before to after the visit is compared between the intervention and control group.

DETAILED DESCRIPTION:
General practices in the Capital Region of Denmark are offered a short educational visit. They are randomized by address to be offered a visit about either proton pump inhibitor (intervention) or another topic (control).

The prescription pattern of each general practice (as seen by their regional registration number [ydernummer]) who receive a visit is investigated.

The change in prescription pattern from before to after the visit is compared between the intervention and control group.

ELIGIBILITY:
Inclusion Criteria:

* General practices in the Capital Region of Denmark, who owns a regional registration number [ydernummer]
* Want a visit
* Have time for a visit within the study period

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Difference in change of number of adult patients with redeemed prescriptions on proton pump inhibitor between asthma-group and placebo-group in a six months period | 6-0 months before and 6-12 months after educational visit
  Difference in change of number of adult patients with redeemed prescriptions on proton pump inhibitor between asthma-group and placebo-group

SECONDARY OUTCOMES:
Difference in change of number of adult patients with redeemed prescriptions on proton pump inhibitor between asthma-group and placebo-group in a one year period | one year before and one year after educational visit
  Difference in change of number of adult patients with redeemed prescriptions on proton pump inhibitor between asthma-group and placebo-group
Difference in change of number of adult patients with redeemed prescriptions on proton pump inhibitor between asthma-group and placebo-group in a one year perioid as interrupted time series analysis | one year before and one year after educational visit
  Difference in change of number of adult patients with redeemed prescriptions on proton pump inhibitor between asthma-group and placebo-group as interrupted time series analysis
Difference in change of number of adult patients with redeemed prescriptions on proton pump inhibitor between asthma-group and placebo-group analyzed by each month in relation to the visit in one year | one year before and one year after educational visit
  Difference in change of number of adult patients with redeemed prescriptions on proton pump inhibitor between asthma-group and placebo-group analyzed by each month in relation to the visit
Difference in change of prescription (DDD) of PPI before and after educational visit in a six months period | 6-0 months before and 6-12 months after educational visit
  Difference in change of defined daily dosages (DDD) of proton pump inhibitor to adult patients between asthma-group and placebo-group
Difference in change of prescription (DDD) of PPI before and after educational visit in one year | one year before and one year after educational visit
  Difference in change of defined daily dosages (DDD) of proton pump inhibitor to adult patients between asthma-group and placebo-group
Difference in change of prescription (DDD) of PPI before and after educational visit in one year as interrupted time series analysis | one year before and one year after educational visit
  Difference in change of defined daily dosages (DDD) of proton pump inhibitor to adult patients between asthma-group and placebo-group as interrupted time series analysis
Difference in change of prescription (DDD) of PPI before and after educational visit in one year for each month | one year before and one year after educational visit
  Difference in change of defined daily dosages (DDD) of proton pump inhibitor to adult patients between asthma-group and placebo-group analyzed by each month in relation to the visit
Difference in change of prescription (DDD) of antacid before and after educational visit in a six months period | 6-0 months before and 6-12 months after educational visit
  Difference in change of defined daily dosages (DDD) of antacid to adult patients between asthma-group and placebo-group
Difference in change of prescription (DDD) of antacid before and after educational visit in one year | one year before and one year after educational visit
  Difference in change of defined daily dosages (DDD) of antacid to adult patients between asthma-group and placebo-group
Difference in change of prescription (DDD) of antacid before and after educational visit in one year as interrupted time series analysis | one year before and one year after educational visit
  Difference in change of defined daily dosages (DDD) of antacid to adult patients between asthma-group and placebo-group as interrupted time series analysis
Difference in change of prescription (DDD) of antacid before and after educational visit in one year for each month | one year before and one year after educational visit
  Difference in change of defined daily dosages (DDD) of antacid to adult patients between asthma-group and placebo-group analyzed by each month in relation to the visit
Difference in change of numbers of big packages of PPI before and after educational visit in a six months period | 6-0 months before and 6-12 months after educational visit
  Difference in change numbers of big packages (90 pcs or more) of PPI in highest dosage strength to adult patients between asthma-group and placebo-group
Difference in change of numbers of big packages of PPI before and after educational visit in one year | one year before and one year after educational visit
  Difference in change numbers of big packages (90 pcs or more) of PPI in highest dosage strength to adult patients between asthma-group and placebo-group
Difference in change of numbers of big packages of PPI before and after educational visit in one year as interrupted time series analysis | one year before and one year after educational visit
  Difference in change numbers of big packages (90 pcs or more) of PPI in highest dosage strength to adult patients between asthma-group and placebo-group as interrupted time series analysis
Difference in change of numbers of big packages of PPI before and after educational visit in one year for each month | one year before and one year after educational visit
  Difference in change numbers of big packages (90 pcs or more) of PPI in highest dosage strength to adult patients between asthma-group and placebo-group analyzed by each month in relation to the visit

CONTACTS AND LOCATIONS:
Overall Officials: Jon tt Andersen, MD, Principal Investigator — University Hospital Bispebjerg and Frederiksberg
Locations (1):
- University Hospital Bispebjerg and Frederiksberg, Copenhagen, Capital Region of Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No